CLINICAL TRIAL: NCT03573570
Title: Reducing Anemia Through Food Fortification at Scale
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Government of Tamil Nadu decided not to proceed with implementation of fortified rice through the Public Distribution (per the original study protocol)
Sponsor: Stanford University (Other)
Collaborators: Government of Tamil Nadu, India (Other); Global Innovation Fund (Other); National AIDS Research Institute (Unknown); King Philanthropies (Unknown)
Responsible Party: Principal Investigator, Grant Miller, Associate Professor, School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-35227
Record Dates: First submitted 2018-05-25; First posted 2018-06-29 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: This project (implementation and accompanying evaluation) will be conducted as a cluster-randomized controlled trial, with baseline and follow-up surveys conducted 12 months apart in the same individuals. In the interim, 110 Treatment Fair Price Shops (FPS) will be assigned randomly to receive rice fortified with iron and other micronutrients, and another 110 Control FPS will be assigned randomly to conventional Public Distribution System (PDS) rice. The control arm therefore represents the status quo and serves as a control group against which any improvements observed in the treatment group will be gauged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 110 Fair Price Shops (FPS) in Chidambaram, Tamil Nadu, India will be assigned randomly to receive rice fortified. Rice will be fortified using Fortified Rice Kernels (FRKs) containing iron, zinc, vitamin A and vitamins B1, B3, B6, B9 and B12. All households receiving rice from the PDS will receive fortified rice instead of conventional PDS rice, and members of households sampled for baseline will have blood samples and demographic surveys taken at a baseline visit, and another visit at 12-15 months after the baseline visit. Because a given FPS only receives rice from a single upstream distributor (godown) it should be straightforward to ensure that fortified rice reaches the appropriate treatment FPS and only those FPS.
  Interventions: Other: Fortified rice kernels
- Control (No Intervention): The control arm, i.e. FPS not a part of the treatment shops, will continue to receive the regular rice supplied by the Public Distribution System (PDS), and members of households sampled for baseline will have blood samples and demographic surveys taken at a baseline visit, and another visit at 12-15 months after the baseline visit. It therefore represents the status quo and serves as a control group against which any improvements observed in the treatment group will be gauged.

INTERVENTIONS:
Other: Fortified rice kernels — The proposed project will leverage the existing state-run public distribution system (PDS) to provide fortified rice through Fair Price Shops (FPS) using a domestically manufactured rice grain (Fortified Rice Kernels: FRK). FRKs are grains made from rice flour, enriched with iron, zinc, Vitamin A, Vitamins B1, B3, B6, B9 and B12, and shaped like a conventional grain of rice. It is mixed into conventional rice in specified ratio of 1:100. The proposed study will be conducted as a cluster-randomized controlled trial, with baseline and follow-up surveys conducted 12-15 months apart. In the interim, 110 Treatment FPS, and all households receiving rice from them, will be randomly assigned to receive fortified rice, and another 110 randomly assigned Control FPS, and the households receiving rice from them, will continue receiving conventional rice and represents the status quo. This study will be conducted in one sub-district of Tamil Nadu with a population of about 1/2 million people.
  Arms: Treatment

SUMMARY:
Anemia is the most common form of malnutrition, affecting approximately 1.6 billion people world-wide. Most commonly caused by iron deficiency, its adverse effects include increased mortality (especially during childbirth), impaired cognitive development among children, chronic fatigue, and reduced lifetime earnings. While iron deficiency is the main cause of anemia worldwide, its etiology is complex and it can also be caused by an insufficient intake of other micronutrients such as Vitamin A, B9, B12 and folate as well as by helminthic infections and malaria.

Research in India and elsewhere has shown that under ideal (controlled) conditions, anemia can be reduced by consumption of iron-fortified food and other micro-nutrients. However, much less is known about the effectiveness of such interventions under actual program conditions on a large scale. This trial proposes to address anemia and other micronutrient deficiencies by providing micronutrient fortified rice through the Public Distribution System (PDS) of Tamil Nadu in a manner that requires no change in behaviour by end-user households and that can feasibly be conducted on a large scale.

This trial is designed as a rigorous cluster-randomized controlled trial with the full collaboration of the government of Tamil Nadu. The trial will follow a randomized cluster design at the Fair Price Shops (FPS) which distribute rice in the Tamil Nadu PDS. Fair Price Shops will be assigned randomly either to the treatment or the control arm, and will either be provided fortified rice for distribution, or the standard, non-fortified rice.

DETAILED DESCRIPTION:
The proposed project will leverage the existing state-run public distribution system (PDS) to provide fortified rice using a domestically manufactured rice grain (Fortified Rice Kernels, or FRK). FRKs are grains made from rice flour, highly enriched with iron and other micronutrients (such as Vitamin A, B9 and Vitamin B12), and shaped like a conventional grain of rice. It is mixed into conventional rice in specified ratios (1g of FRK 100g of conventional rice) and is almost indistinguishable from conventional rice in appearance and taste. For this study, rice will be fortified using FRKs containing iron, zinc, vitamin A and vitamins B1, B3, B6, B9 and B12.

The Tamil Nadu PDS already provides up to 20 kilograms of rice at no cost to all households in the state, with an additional 15 kilograms to households identified as particularly poor. This is done through a widespread network of Fair Price Shops (FPS). The proposed study (implementation and accompanying evaluation) will be conducted as a cluster-randomized controlled trial, with baseline and follow-up surveys conducted 12-15 months apart. In the interim, 110 Treatment FPS will be randomly assigned to receive fortified rice, and another 110 randomly assigned Control FPS will continue receiving conventional rice. The investigators plan to conduct the study in one sub-district of Tamil Nadu with a population of about 1/2 million people.

In a cluster, the study team will randomly select 40 households to participate in the baseline and followup surveys and household members meeting the eligibility criteria, i.e. women between 12 and 40 years and children between 6 and 59 months, will be enrolled. These surveys will collect information about dietary patterns and socioeconomic status, and importantly, will also collect objectively measured health indicators (biomarkers and anthropometric measures), to test directly for anemia and micronutrient deficiencies.

To implement the intervention, the Government pre-existing PDS system, will be used. Every household in Tamil Nadu has a card that entitles it monthly to a pre-specified quantity of rice (and other goods) from a specific location that belongs to a network of so called Fair Price Shops (FPS). These FPS in turn receive rice from government-run warehouses (called godowns) where rice is delivered from a central procurement system and then bagged.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age group of 6 months to 5 years
* Women in the age group of 12 to 40 years

Exclusion Criteria:

* None

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin level from baseline to endline using Rapid Diagnostic Tests (RDT) | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Rapid Diagnostic Tests (RDT), using Hemocue machine, will be used to measure Hemoglobin concentrations in 40 women and 40 children tested in each FPS catchment area (total sample size 17600 women and children). Hemoglobin (Hb) will be tested with the HemoCue analyzer, a portable, accurate system for measuring Hb. Hb measures will be used to calculate prevalence of anemia among the target population of women and young children. The test requires less than 0.5 ml of blood and delivers results in approximately 15 minutes.
Change in hemoglobin level from baseline to endline using DBS | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Hemoglobin (Hb) will also be measured separately in a sub-sample of individuals (10 children and 10 women per FPS) using Dried Blood Spots (DBS) that will be transported to a lab for analysis. It will take up to 15 minutes for each respondent.
Change in Transferrin Receptor (TfR) level from baseline to endline using DBS | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Transferrin Receptor (TfR) will also be measured separately in a sub-sample of individuals (10 children and 10 women per FPS) using Dried Blood Spots (DBS) that will be transported to a lab for analysis. TfR is a good indicator of iron stores in the body, and this marker is expected to improve following food fortification. C-Reactive Protein (CRP) will also be measured. CRP is useful both to detect the presence of inflammation and to identify cases where measured TfR is likely to give a biased account of iron stores, given that TfR becomes elevated in the presence of acute and sometimes chronic infections; thus, TfR will be corrected for inflammation using CRP. It will take up to 15 minutes for each respondent.
Change in anemia measured by RDT (Hemocue machine) and DBS from baseline to endline | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Anemia measured by RDT (Hemocue machine) and DBS: Hb measured from RDT, i.e. Hemocue machine, and DBS will further be categorized to estimate the prevalence of anemia among the study population using established Hb thresholds. Based on the WHO classification, the following thresholds will be considered:
  For children aged 6 to 59 months:
  * No anemia: Hb >= 11 g/dL
  * Mild anemia: 10 < Hb < 10.9 g/dL
  * Moderate anemia: 7 < Hb < 9.9 g/dL
  * Severe anemia: Hb < 7 g/dL
  For non-pregnant women aged 12 years and above:
  * No anemia: Hb >= 12 g/dL
  * Mild anemia: 11 < Hb < 11.9 g/dL
  * Moderate anemia: 8 < Hb < 10.9 g/dL
  * Severe anemia: Hb < 8 g/dL
  For pregnant women aged 12 years and above:
  * No anemia: Hb >= 11 g/dL
  * Mild anemia: 10 < Hb < 10.9 g/dL
  * Moderate anemia: 7 < Hb < 9.9 g/dL
  * Severe anemia: Hb < 7 g/dL

SECONDARY OUTCOMES:
Change in height from baseline to endline | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Height will be measured for all study participants (children that are 6 months and older, and women between the ages of 12 and 40 years) at baseline and endline. This will take up to 10 minutes.
Change in weight from baseline to endline | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Weight will be measured for all study participants (children that are 6 months and older, and women between the ages of 12 and 40 years) at baseline and endline. This will take up to 10 minutes.
Change in productivity from baseline to endline | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Employment status, hours worked, productivity, and earnings will be measured for working age adults at baseline and endline. This will take approximately 10 minutes.
Change in cognitive outcomes for children from baseline to endline | This will be assessed at baseline and at endline after 12-15 months of intervention.
  Cognitive outcomes for children using Development Milestones Checklist and Wechsler Preschool and Primary Scale of Intelligence instruments, as well as school enrollment and attendance data for older children will be measured. This will take approximately 30 minutes to administer.

CONTACTS AND LOCATIONS:
Overall Officials: Norman G Miller, PhD, Principal Investigator — Stanford University; Aprajit Mahajan, PhD, Principal Investigator — University of California, Berkeley; Alessandro Tarozzi, PhD, Principal Investigator — Universitat Pompeu Fabra; Reynaldo Martorell, PhD, Principal Investigator — Emory University
Locations (1):
- Institute for Financial Management and Research (IFMR) and Cuddalore district, Tamil Nadu, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be shared upon successful publication of the main paper from the project.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At the time of publication of the main paper from the project (and in perpetuity afterwards)
Access Criteria: All shared materials will be publicly available i.e. there are no other access criteria